CLINICAL TRIAL: NCT05708625
Title: Efficacy of Intralesional Voriconazole Versus Intralesional Cryotherapy Versus Intralesional Sodium Stibogluconate Versus Oral Doxycycline in the Treatment of Acute Cutaneous Leishmaniasis
Brief Title: Intralesional Voriconazole, or Intralesional Cryotherapy, or Oral Doxycycline in the Treatment of Cutaneous Leishmaniasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hagar Nofal, Clinical Professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#8095/3-10-2021
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Voriconazole; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intralesional Sodium stibogluconate (Active Comparator): Patients will receive intralesional infiltration of (SSG) at a dose of 50 mg/0.5 ml (0.2-0.4ml) maximum dose per session 1-3 ml. Sessions will be held once weekly for a maximum of 6 weeks.
  Interventions: Drug: Intralesional Sodium stibogluconate
- intralesional Cryotherapy (Experimental): Patients will be treated with intralesional Cryotherapy. Sessions will be held every two weeks till complete cure or a maximum of 6 sessions
  Interventions: Procedure: Intralesional Cryotherapy
- Intralesional Voriconazole (Experimental): Patients will be treated with intralesional Voriconazole weekly till complete cure or a maximum of 6 sessions
  Interventions: Drug: Intralesional Voriconazole
- Oral doxycycline (Experimental): Patients will be treated with oral doxycycline, 200 mg daily, until complete cure or a maximum of 6 weeks
  Interventions: Drug: Oral doxycycline

INTERVENTIONS:
Drug: Intralesional Sodium stibogluconate — Sessions will be held once weekly for a maximum of 6 weeks
  Other Names: SSG
  Arms: Intralesional Sodium stibogluconate
Procedure: Intralesional Cryotherapy — Intralesional Cryotherapy. Sessions will be held every two weeks
  Arms: intralesional Cryotherapy
Drug: Intralesional Voriconazole — Weekly intralesional Voriconazole
  Other Names: Vfend
  Arms: Intralesional Voriconazole
Drug: Oral doxycycline — 200 mg daily for 6 weeks or till complete cure
  Arms: Oral doxycycline

SUMMARY:
Leishmaniasis is a vector-borne disease caused by obligate, intracellular protozoa of the genus Leishmania and transmitted by phlebotomine sandflies. It is found mostly in tropical and subtropical areas then it has spread into southern Europe. Increased international travel and immigration have led to an increased diagnosis of leishmaniasis cases in nonendemic areas (Kollipara et al., 2016). Foci of CL, caused by L. ma¬jor, occur in Afghanistan, Egypt, Iran, Iraq, Jordan, Libya, Morocco, Palestine, Pakistan, Saudi Arabia, Sudan, Syria, Tunisia, and Yemen. Many researchers have studied leishmaniasis in the endemic northern African countries, e.g., Morocco, Algeria, Tunisia, Egypt, and Libya. One of the established endemic leishmaniasis Libyan provinces is Al-jabal Al-gharbi province, where CL comprises a major parasitic health problem (Abdellatif et al., 2013).To evaluate the efficacy of intralesional cryotherapy, intralesional Voriconazole, and oral doxycycline in the treatment of cutaneous leishmaniasis compared to the conventional treatment (intralesional SSG).

DETAILED DESCRIPTION:
* Cutaneous leishmaniasis is a prevalent parasitic infection in northern Africa. In Egypt, CL cases are detected mainly in eastern governorates including Sinai. Cutaneous leishmaniasis represent a socioeconomic burden on the affected communities.
* Available treatment options are expensive and associated with systemic toxicity. There are alarming reports of emerging resistance against the currently in use therapeutics. Comparative controlled trials for the effective and the least harmful treatment modalities are lacking.
* Up to our knowledge this is the first study investigating the effectiveness of intralesional Voriconazole and intralesional cryotherapy in the treatment of cutaneous leishmaniasis

So in this study the following objectives are being aimed:

1. To evaluate the effectiveness and safety of intralesional Voriconazole comparing it to the intralesional SSG in patients with CL.
2. To evaluate the effectiveness and safety of intralesional cryotherapy comparing it to the intralesional SSG in patients with CL.
3. To evaluate the effectiveness and safety of Oral doxycycline comparing it to the intralesional SSG in patients with CL.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be willing to sign informed consent, for patients younger than 18 years old, parents or guardians will sign an informed consent.

  1. Patients clinically diagnosed with cutaneous leishmaniasis and confirmed using parasitological Giemsa-stained direct smears.
  2. Acute lesions of less than 12-week duration to exclude any possibility of natural self-healing of the lesions during follow-up.
  3. Both sexes.
  4. Age: > 12 years old.

Exclusion Criteria:

* • Pregnancy and lactation.

  * Patients < 12 years old.
  * Patients with negative Giemsa stained direct smears.
  * Patients with concomitant renal or liver impairment, congestive heart failure, uncontrolled diabetes mellitus, peripheral neuropathy, poor peripheral circulation, and prolonged corticosteroid therapy.
  * Patients with lesions of more than 12 weeks duration.
  * Patients with lesions > 5cm2
  * History of anti-Leishmania therapy in the last 3 months.
  * For the intralesional groups the presence of > 5 lesions.
  * Lesions in the perimeter (< 2 cm) of mucosal areas e.g. eyes, nose, mouth, or genitals.
  * Patients with known hypersensitivity or allergy to the assigned drugs.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response to treatment | 6 weeks
  The responses will be graded by an investigator who don't perform the injections. The clinical response will be graded based on the improvement percentage of the lesion in terms of size, erythema, inflammation, edema and ulcer re-epithelialization

SECONDARY OUTCOMES:
Persistence of clinical response | 12 week post treatment termination
  Persistence of clinical response at the end of follow-up period
Patient compliance | 6 weeks
  The percentage of patients continued the study in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Nofal, Dr, Principal Investigator — Zagazig University
Locations (1):
- Dermatology department, Gharyan University Hospitals, Medical College, Gharyan University, Gharyan, Select Region, Libya

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Akulinina IK, Berechikidze IA, Larina SN, Sakharova TV, Degtyarevskaya TY, Romanelli M. Effectiveness of doxycycline for the treatment of zoonotic cutaneous leishmaniasis in vivo. Parasitology. 2021 Mar;148(3):361-365. doi: 10.1017/S0031182020002152. Epub 2020 Nov 16. PMID 33190654
- [Background] Asilian A, Sadeghinia A, Faghihi G, Momeni A. Comparative study of the efficacy of combined cryotherapy and intralesional meglumine antimoniate (Glucantime) vs. cryotherapy and intralesional meglumine antimoniate (Glucantime) alone for the treatment of cutaneous leishmaniasis. Int J Dermatol. 2004 Apr;43(4):281-3. doi: 10.1111/j.1365-4632.2004.02002.x. PMID 15090013
- [Background] Bahrami S, Oryan A, Bemani E. Efficacy of amiodarone and voriconazole combination therapy in cutaneous leishmaniasis in the mice experimentally infected with Leishmania major. J Infect Chemother. 2021 Jul;27(7):984-990. doi: 10.1016/j.jiac.2021.02.011. Epub 2021 Feb 23. PMID 33637428
- [Background] Daie Parizi MH, Karvar M, Sharifi I, Bahrampour A, Heshmat Khah A, Rahnama Z, Baziar Z, Amiri R. The topical treatment of anthroponotic cutaneous leishmaniasis with the tincture of thioxolone plus benzoxonium chloride (Thio-Ben) along with cryotherapy: a single-blind randomized clinical trial. Dermatol Ther. 2015 May-Jun;28(3):140-6. doi: 10.1111/dth.12229. Epub 2015 Apr 6. PMID 25847678
- [Background] Soto J, Rojas E, Guzman M, Verduguez A, Nena W, Maldonado M, Cruz M, Gracia L, Villarroel D, Alavi I, Toledo J, Berman J. Intralesional antimony for single lesions of bolivian cutaneous leishmaniasis. Clin Infect Dis. 2013 May;56(9):1255-60. doi: 10.1093/cid/cit049. Epub 2013 Feb 6. PMID 23390069